CLINICAL TRIAL: NCT05273424
Title: Clinical Outcomes of Chronic Kidney Disease Patients on Hemodialysis in Brazil: A Prospective Cohort Study
Brief Title: Clinical Outcomes of Hemodialysis in Brazil (COHEBRA): a Prospective Cohort Study
Acronym: COHEBRA
Status: Enrolling by invitation | Type: Observational
Sponsor: Catholic University of Pelotas (Other)
Collaborators: Federal University of Pelotas (Other)
Responsible Party: Principal Investigator, Maristela Bohlke, Professor, Catholic University of Pelotas
Other Study IDs: COHEBRA
Record Dates: First submitted 2021-10-18; First posted 2022-03-10 (Actual); Last update posted 2022-03-10 (Actual); Status verified 2022-02

CONDITIONS: Chronic Kidney Diseases; Hemodialysis Complication
MeSH Terms: conditions — Renal Insufficiency, Chronic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- no groups: A cohort of CKD patients on hemodialysis

SUMMARY:
Introduction: Chronic kidney disease (CKD) is characterized by progressive decrease in glomerular filtration rate (GFR), eventually reaching the end-stage renal disease (ESRD) requiring renal replacement therapy (RRT). The decrease in GFR is associated with a linear increase in cardiovascular mortality. Dysfunction of the autonomic nervous system (ANS) has been well documented in patients with CKD, especially in people with ESRD. The renal ischemia causes both the excessive activation of the renin-angiotensin-aldosterone system (RAAS) by increasing renin release, as sympathetic ANS, through the afferent sympathetic nerves. The overactivated RAAS and sympathetic SNA feedback each other, which contributes to cardiovascular disease (CVD) in CKD. Despite the involvement of these systems in the pathogenesis of CVD in CKD, drugs that block the RAAS or sympathetic SNA have shown heterogeneous effects in CVD in this population. A potential explanation is the genetic heterogeneity, such as the polymorphism in the gene for angiotensin converting enzyme (ACE).In addition, the inflammatory process associated with CKD is regarded as central player in the general degenerative changes backing CKD on HD shorter survival, which in many aspects is like accelerated aging. Skeletal muscles are also affected in a pattern like aging sarcopenia, with loss of function and mass. Objectives: to evaluate the impact of ECA gene polymorphism, HRV, body composition, functional capacity, muscle strength, inflammatory factors and other potential predictors on the survival of patients with CKD treated by HD in a single center in southern Brazil. Methodology: Prospective cohort study. The sample will consist of adult patients with CKD on HD longer than 90 days. Sociodemographic and clinical data is collected from clinical records. HRV analysis is performed using a Micromed@ electrocardiogram device® with a recording of the standard deviation of all normal intervals (SDNN), square root of the mean of the squares of the differences between consecutive intervals (RMSSD), low frequency band (LF) and high frequency (HF) after a midweek HD session. The polymorphism of the ECA gene was evaluated by polymerase chain reaction method in peripheral blood DNA sample. Muscle quality and thickness has been obtained by ultrasound. Functional capacity by 6-minute walking test and muscle strength by dynamometer. The data will be analyzed using Stata 15.0 statistical package.

DETAILED DESCRIPTION:
Evaluation of HRV. HRV measurement was performed using an electrocardiographic device (Wincardio@, Micromed). The registry was acquired for 20 min before, in the second hour, and immediately after a midweek HD session. Patients were in a supine position and breathed normally during the recording. Patients with unstable patterns of breath had their HRV recording postponed. The electrocardiographic device transmitted the R-R interval record to digital storage, which was subsequently analyzed in the time and frequency domains of HRV through CardioSeries@ 2.4 software. In the time domain, RMSSD and SDNN were acquired. In the frequency domain analysis, a tachogram was interpolated in a frequency of 4 Hertz and divided into periods of 256 points with 50% overlap. These signals were submitted to spectral analysis by fast Fourier transformation to obtain the total power of the spectrum. The LF band, representing sympathetic modulation, was between 0.02 and 0.15 Hz. The HF band, attributed to parasympathetic modulation, was between 0.15 and 0.40 Hz.

ACE gene typing. Blood samples were drawn and centrifugated. The leukocyte supernatant pellet was extracted and stored. ACE polymorphism was typed by PCR for DD, ID, and II genotypes. It used the following specific primers for DNA amplification: sense 5=-CTGGAGACCACTCCCATCCTTTCT-3= and antisense 5= GATGTGGCCATCACATTCGTAGA- 3=. Through these primers, it was possible to detect allele deletion and insertion. A confirmatory PCR was done for all samples with the DD genotype to increase the specificity of the genotyping using a pair of specific primers for insertions, i.e., an allele I amplifier. These primers were as follows: sense 5=-TGGGACCACAGCGCCCGCCACTAC-3= and antisense 5=-TCGCCAGCCCTACCATGCCCATAA-3=. The temperature protocol was programed in the thermocycler beginning at 95°C for 5 min and then 40 cycles of denaturation at 95°C for 45 s, annealing at 54°C for 1 min, and extension at 72°C for 30 s each and then at 5 min at 72°C to finish uncompleted chains.

Hydration status assessment. The patient's hydration status was evaluated before and after (up to 20 min) the studied HD session using a Body Composition Monitor (Fresenius), which uses multifrequency bioimpedance spectroscopy to determine the electrical resistances of total body water and extracellular water. Electrodes were attached to the hand and feet opposite to vascular access, with the patient in a supine position, and the measurement was done and stored in a digital format and analyzed with the Fluid Management Tool. The results were provided as overhydration (in liters), which represents the excess of water above reference levels according to the patient's sex and age.

Muscle thickness and echo intensity by ultrasound Patients were evaluated after one midweek dialysis session. They initially were instructed to stand with the legs and ~20 cm apart. The length of right thigh was measured from the superior iliac spine to the proximal border of the patella. Right and left circumferences were assessed at the midpoint of the thighs. At the same level on the anterior face of the thighs, skin was marked with a water-resistant pen. The quadriceps thickness was measured with the probe over these points, perpendicular to the long axis of the limb (cross-sectional image) and captured after proper visualization of the bone surface. The image was stored in device's hard disk for each of the two sites.

The images were analyzed later using the software ImageJ (National Institute of Health, USA, version 1.37) for both muscle thickness and echo intensity (EI). The thickness was measured as the perpendicular distance between the point just above the apex of the femur surface and the point just below the rectus femoris' superficial fascia obtained using the same software with the length function. The measurements were registered in millimeters and posteriorly converted to centimeters.

The EI analysis was performed after the selection of a record region that includes as much muscle as possible while avoiding surrounding fascia. The EI was then calculated from the selected region with gray-scale analysis using the standard histogram function and expressed in values between 0 and 255 (0 = black; 255 = white) (Radaelli et al., 2013; Wilhelm et al., 2014).

Functional capacity - six-minute walking test Functional capacity was measured using the 6-minute walk test (6MWT). This test is a submaximal effort test, affordable and easy to perform, in addition to be well established as representative of functional capacity in frail subjects. The 6-minute walk test shows a good correlation with the maximal oxygen uptake measure. The result of 6MWT in meters was multiplied by 100 and divided by the predicted distance for age. The result (percent of predicted distance walked by age) was used in analysis.

Muscle strength assessment Evaluation of muscle strength was performed using the static strength test of the legs, using a Crown® (Oswaldo Filizola Industry, São Paulo, Brazil) dynamometer. The measurement was repeated after a 1-minute interval. The mean of the two measurements was used in the analysis.

ELIGIBILITY:
Inclusion Criteria:

* chronic kidney disease
* hemodialysis treatment for longer than 90 days

Exclusion Criteria:

* According to outcomes evaluated

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult chronic kidney disease on hemodialysis
Sampling Method: Non-Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-06-01 (Actual); Primary Completion 2021-06-01 (Actual); Study Completion 2027-06-01 (Estimated)

PRIMARY OUTCOMES:
survival | ten years
  survival time

SECONDARY OUTCOMES:
hospital admission | ten years
  hospital admission rate

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital Universitário São Francisco de Paula, Pelotas, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided